CLINICAL TRIAL: NCT06840106
Title: Effectiveness and Safety of Nasal Herbal Steam Therapy for Post-extubation Respiratory Events : Pragmatic Randomized Controlled, Parallel Grouped Study
Brief Title: Nasal Steam Therapy for Post-extubation Respiratory Events
Acronym: PURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilsan Cha hospital (Other)
Responsible Party: Principal Investigator, Jee Young Lee, Assistant professor, Ilsan Cha hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICICC-CT-24-01
Record Dates: First submitted 2025-01-21; First posted 2025-02-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Thyroid Cancer; Intubation
Keywords: thyroid cancer; post-extubaton; upper respiratory event
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Nasal steam therapy is performed once a every other day for a total of 3three times. The steam inhalation stimulates the acupoints of bilateral LI20, EX-HN8, and EX-HN9
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and the statistician will be blinded to evaluate the efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal Steam therapy strategy (Experimental): Nasal steam therapy is performed once a every other day for a total of 3three times. The steam inhalation stimulates the acupoints of bilateral LI20, EX-HN8, and EX-HN9
  Interventions: Procedure: Nasal steam therapy
- Routine management strategy (Active Comparator): This study is a practical clinical study, and the selection of drugs and other treatment methods will be based on the doctor's clinical judgment regarding the patient's symptoms, degree of improvement, etc. Drug administration or patient education will be implemented according to symptoms. Depending on the patient's symptoms and degree of improvement, the clinician may utilize all drugs currently used in clinical practice to improve upper respiratory symptoms, if necessary. All drugs that fall under the Anatomical Therapeutic Chemical Classification System (ATC) codes of non-disease treatment (R01), throat disease treatment (R02), lung disease or expectorant (R03, R05), and other respiratory organ drugs (R06, R07) and other drugs that clinicians orally administer in current clinical practice for the purpose of improving upper respiratory symptoms will be collected.
  Interventions: Procedure: Routine management strategy

INTERVENTIONS:
Procedure: Nasal steam therapy — Nasal steam therapy is performed once a every other day for a total of 3three times. The steam inhalation stimulates the acupoints of bilateral LI20, EX-HN8, and EX-HN9
  Arms: Nasal Steam therapy strategy
Procedure: Routine management strategy — Depending on the patient's symptoms and degree of improvement, the clinician may utilize all drugs currently used in clinical practice to improve upper respiratory symptoms, if necessary. All drugs that fall under the Anatomical Therapeutic Chemical Classification System (ATC) codes of non-disease treatment (R01), throat disease treatment (R02), lung disease or expectorant (R03, R05), and other respiratory organ drugs (R06, R07) and other drugs. The usage and dosage should be within the range of the current clinical guidelines.
  Arms: Routine management strategy

SUMMARY:
The effect of symptom improvement of nasal steam strategy compared to routine management strategy for upper respiratory symptoms occurring after endotracheal intubation in patients aged 19 years or older who underwent surgical removal under anesthesia requiring endotracheal intubation was evaluated by the difference in the results of Wisconsin Upper Respiratory Symptom Survey

DETAILED DESCRIPTION:
This study aims to confirm the comparative effectiveness of nasal steam therapy by conducting a practical randomized controlled clinical trial comparing 66 patients complaining of upper respiratory symptoms with patients treated with a nasal steam therapy strategy (33 patients) and patients treated with a routine management strategy (33 patients).

This study is a practical clinical study, and only randomly assigns patients to two groups: nasal steam therapy strategy and routine management strategy. The specific treatment method used is not determined in advance. The specific treatment is performed according to the clinical judgment according to the patient's condition. All treatment methods used during the study are recorded in the case report and compared.

The treatment will be administered for a total of 5 days, and drug treatment may not be discontinued after the study period at the clinician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 to 69 years

  * Those who underwent surgical removal of the thyroid gland under endotracheal intubation due to a thyroid tumor

    * American Society of Anesthesiologists (ASA) status I or II

      * Those who developed upper respiratory symptoms after surgery ⑤ Voluntarily decided to participate in this clinical trial and signed the informed consent form

Exclusion criteria:

* Those diagnosed with symptomatic gastroesophageal reflux disease

  * Chronic cough lasting for more than 3 months prior to surgery, including bronchial asthma and chronic obstructive pulmonary disease (COPD)

    * Those who developed other respiratory infections within the past month ④ Those who are taking or are required to take other medications that may interfere with the interpretation of the treatment effect or results

      * Those who are scheduled to undergo additional major treatments such as reoperation, chemotherapy, and radiotherapy during the clinical trial period ⑥ Pregnant women, breastfeeding women, and those who plan to become pregnant during the study period ⑦ Others who are expected to have difficulty complying with the treatment, visits, and questionnaires stipulated in this protocol at the discretion of the medical staff

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Wisconsin upper respiratory symptom survey-24, WURSS-24 | From enrollment to the end of treatment at Day 8, and follow up visit at Day 15
  WURSS is a questionnaire mainly used to evaluate symptoms of acute upper respiratory tract infection, and is divided into WURSS-11, WURSS-21, WURSS-24, WURSS-44, and WURSS-Kids versions. In this study, WURSS-24 will be used to evaluate the degree of daily symptom improvement by dividing it into items of symptoms, quality of life, and overall satisfaction, and 24 questions on a 7-point Likert scale. The most severe level is evaluated as 7 points, the least level as 1 point, and in the case of symptoms and quality of life that may be lost, 0 points are additionally recorded when the symptoms are lost.

SECONDARY OUTCOMES:
Incidence and severity of cough | Day 1, Day 4, Day 8, Day 15
  * The number of times the participant experienced coughing during the day will be recorded.
  * The degree of discomfort in your daily life due to coughing will be assessed using the numeric rating scale (NRS). On the NRS, the patient selects a number from 0 to 10 that best represents their current level of discomfort (0 being no discomfort, 10 being the worst discomfort imaginable).
Thyroid cancer-Quality of Life (ThyCa-QoL) | Day 1, Day 4, Day 8, Day 15
  - THYCA-QoL is a health-related quality of life questionnaire developed for thyroid cancer and thyroid cancer survivors. It was developed using methodologically proven standard guidelines and is a validated questionnaire that can improve symptoms, treatment, aftercare, and disease experience of thyroid cancer survivors.

CONTACTS AND LOCATIONS:
Locations (1):
- Ilsan Cha Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This study is part of a national project and data will be provided based on the decision of the Korea Health Industry Development Institute under the Ministry of Health and Welfare.